CLINICAL TRIAL: NCT03586960
Title: Use of a Novel Device for Stretch Relaxation During Mohs Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Silver Falls Dermatology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB18-025
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Tissue Expander Disorder; Stress Strain Curve; Tissue Expansion; Mohs Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental Group (Experimental): Peak tension will be measured with a calibrated force gauge (Series 3 Digital Force Gauge; Mark-10 Corporation; Copiague, NY) until the wound edges touch. A clamp will be used to secure the sutures on top of the device between measurements. At each time point (5, 10 and 30 minutes), the clamps will be loosened and the wound allowed to relax. Photographs and measurements will be taken to document the wound size after stress-reduction. The suture will be re-tensioned while measurements of peak tension (as outlined above) are recorded with the force gauge.
  Interventions: Device: Peak Force Measurement

INTERVENTIONS:
Device: Peak Force Measurement — Force will be measured at 5,10, and 30 minutes

SUMMARY:
Closure of cutaneous defects is associated with many common and serious problems. For example, Mohs surgery involves the removal of skin and other soft tissues that have been proven to be infiltrated with cancer. Iterative stages of Mohs are processed and examined microscopically for residual tumor. Using specialized mapping, the surgeon can effectively achieve a high cure rate and minimize removal of unaffected tissue. This process usually takes a total of 2-3 hours, since the patient waits while the tissue is being processed, and complete clearance of margins can take multiple stages. In many cases, a cutaneous defect is produced of significant size. In certain areas of high tension, such as scalp and lower leg, this mandates either a lengthy course of wound care or that the surgeon perform a graft or flap. In many cases, performance of a graft is undesirable due to lack of vascularity to support graft survival. Creation of flaps involves incision and undermining of large areas of tissue in order to achieve wound closure. There is a current need for alternatives to graft and flaps in these locations.

Human skin has biomechanical properties that can be harnessed to facilitate closure of larger wounds. Stress-relaxation refers to the natural relaxation exhibited by skin put under a given amount of tension (stress) over time. After a period of stress, the force required to close the wound is reduced. In a porcine skin wound model, there is a 40-60% reduction in stress after twenty minutes of stretch relaxation.

There are several classic methods of delivering this stretch to skin intraoperatively. Most simply, a towel clamp can be used to bring edges together. However, the clamp, which is a sharp stainless steel instrument, can damage tissues. There are also commercial devices such as TopClosure. However, this device is intended for very large wounds with side plates that must be sutured or stapled to patient skin.

The SUTUREGARD device presents a simple method to provide stress to a wound but not damage tissue. The SUTUREGARD device results in significantly lower pressure on the skin when compared with traditional sutures and creates a much greater volume of wound eversion than is possible with a traditional suturing method. Engineering tests performed at OSU showed that a given simple interrupted suture will exert about 30% less pressure on the skin when used performed with the device compared to without the device. With this protection, this creates the corollary that a suture could be safely tied to a greater force with the device than without. In animal testing, the device has been used on porcine wounds for up to 6 weeks, where it showed superior histologic tolerability over traditional sutures.

The investigators have used the device to provide stress-relaxation within our clinic over the past several months and have seen reductions in wound width of about 30% with retention of the device for 30-60 minutes. Wounds exhibit significantly more reduction in width with overnight use. Unlike traditional retention sutures, which damage the skin, the skin appears normal with retention of the device for up to 2 days in our patients. Furthermore, all wounds that have been stress-relaxed with the device have healed without complication.

The investigators plan to study the stress-relaxation created by use of a SUTUREGARD device applied to cutaneous defects for a specified time periods (30, 60 and 90 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Any wound that cannot be reapproximated upon tumor removal (These locations are often on the lower leg and scalp.)
* Age over 18 years
* Intact skin surrounding wound for at least 2.5 cm

Exclusion Criteria:

* Active infection
* Systemically unstable or unwell patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Direct measurements of wound dimensions at each timepoint | 5 minutes
  Measurements will be taken at each time point of wound size
Direct measurements of wound dimensions at each timepoint | 10 minutes
  Measurements will be taken at each time point of wound size
Direct measurements of wound dimensions at each timepoint | 30 minutes
  Measurements will be taken at each time point of wound size

CONTACTS AND LOCATIONS:
Locations (1):
- Silver Falls Dermtology, Salem, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saqib NU, Domenick N, Cho JS, Marone L, Leers S, Makaroun MS, Chaer RA. Predictors and outcomes of restenosis following tibial artery endovascular interventions for critical limb ischemia. J Vasc Surg. 2013 Mar;57(3):692-9. doi: 10.1016/j.jvs.2012.08.115. Epub 2013 Jan 23. PMID 23351646
- [Background] Townsend KL, Akeroyd J, Russell DS, Kruzic JJ, Robertson BL, Lear W. Comparing the Tolerability of a Novel Wound Closure Device Using a Porcine Wound Model. Adv Wound Care (New Rochelle). 2018 Jun 1;7(6):177-184. doi: 10.1089/wound.2017.0777. PMID 29892494
- [Background] Topaz M, Carmel NN, Topaz G, Li M, Li YZ. Stress-relaxation and tension relief system for immediate primary closure of large and huge soft tissue defects: an old-new concept: new concept for direct closure of large defects. Medicine (Baltimore). 2014 Dec;93(28):e234. doi: 10.1097/MD.0000000000000234. PMID 25526444
- [Result] Hussain SH, Limthongkul B, Humphreys TR. The biomechanical properties of the skin. Dermatol Surg. 2013 Feb;39(2):193-203. doi: 10.1111/dsu.12095. Epub 2013 Jan 25. PMID 23350638